CLINICAL TRIAL: NCT03203395
Title: Screening for Depression and Anxiety in Patients With Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Extrastiftelsen (Other); LHL - The Norwegian Heart and Lung Patient Organization (Unknown)
Responsible Party: Principal Investigator, Torkil Berge, Academic Development Counselor, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016/16558 (PVO); 2016/16558 (Other: The Data Protection Officer (Personvernombudet))
Record Dates: First submitted 2017-06-23; First posted 2017-06-29 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Depression; Depressive Symptoms; Depressive Disorder; Anxiety; Anxiety Disorders; Panic Attacks; Heart Diseases; Collaboration
Keywords: Depression; Anxiety; Panic Attacks; Collaborative Care; Heart disease and depression; Heart disease and anxiety; Heart disease and panic attacks
MeSH Terms: conditions — Depression; Depressive Disorder; Anxiety Disorders; Panic Disorder; Heart Diseases | interventions — Mass Screening; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart patients (Experimental): Screening and counselling
  Interventions: Behavioral: Screening and counselling

INTERVENTIONS:
Behavioral: Screening and counselling — Screening for symptoms of depression and anxiety in heart patients, giving advice for prevention and managing of such symptoms and stimulating collaborative care between the hospital and the general practitioner.

SUMMARY:
Depression is a risk factor for morbidity and mortality in patients with heart disease, and has a negative impact on quality of life, work capacity and treatment adherence. Screening for depression among heart patients are therefore recommended by the Norwegian Health Authorities. Also, symptoms of anxiety may negatively affect rehabilitation due to e.g. fear of physical activity and excessive worry. Patients currently receiving treatment for heart disease at Diakonhjemmet Hospital will be screened for symptoms of depression and anxiety. If such symptoms are detected, patients will be offered a counselling session with a clinical psychologist. Further, routines for collaborative communication between clinical psychologist, cardiologist and the patient's general physician will be emphasized.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years under treatment for myocardial infarction, heart failure, tachyarrhythmia and/or valvular heart disease at the Department of Internal Medicine, Diakonhjemmet Hospital.

Exclusion Criteria:

* Unable to provide informed consent.
* Unable to read and/or understand Norwegian.
* Unable to complete a survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Detection of symptoms of depression, anxiety and/or recent panic attack in heart patients. | 15 minutes
  All patients included in the study will be screened for symptoms of depression, anxiety and recent panic attack by filling out a survey consisting of questions from the Patient Health Questionnaire-2 (PHQ-2), the Generalized Anxiety Disorder Scale-2 (GAD-2) and a question about whether they experienced a panic attack in the last four weeks. Cut-off is set to a score of ≥ 2 on PHQ-2 and/or GAD-2 and/or a positive answer on the question about panic attack.
Detection of patients with or at risk for depression and/or anxiety disorders. | 1 hour
  Patients who screened positive for symptoms of depression, anxiety and/or panic attack will be asked to complete the Hospital Anxiety and Depression Scale (HADS). Patients with a HADS score of ≥ 4 will be offered a counselling session with a clinical psychologist.
Implementation of counselling for treatment and prevention of depression and anxiety disorders in heart patients. | 1-2 hours
  Patients with a HADS score of ≥ 4 will be offered a counselling session with a clinical psychologist aimed to treat and prevent depression and anxiety disorders in heart patients.

CONTACTS AND LOCATIONS:
Overall Officials: Torkil Berge, Psychologist, Principal Investigator — Department of Psychiatry, Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No